CLINICAL TRIAL: NCT01468818
Title: A Pilot Study of the Administration of Young Tumor Infiltrating Lymphocytes Following a Non-Myeloablative Lymphocyte Depleting Chemotherapy Regimen in Metastatic Melanoma
Brief Title: Immunotherapy Using Tumor Infiltrating Lymphocytes for Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed prematurely due to slow and insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110260; 11-C-0260
Record Dates: First submitted 2011-10-06; First posted 2011-11-10 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Metastatic Melanoma; Skin Cancer
Keywords: Metastatic Melanoma; Adoptive Cell Therapy; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunotherapy for Metastatic Melanoma (Experimental): Patients will receive non-myeloablative lymphodepleting preparative regimen cons
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Young Tumor Infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
Drug: Fludarabine — Fludarabine 25 mg/m2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
Biological: Young Tumor Infiltrating Lymphocytes (TIL) — Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of young TIL. On day 0, cells (1x10e9 to 2x10e11) will be infused intravenously (i.v.) on the Patient Care Unit over 20 to 30 minutes (between one and four days after the last dose of fludarabine).

SUMMARY:
Background:

* The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy that involves taking white blood cells from patients' tumors, growing them in the laboratory in large numbers, and then giving the cells back to the patient with aldesleukin (IL-2) a drug that keeps the white blood cells active. These cells are called Tumor Infiltrating Lymphocytes, or TIL and we have given this type of treatment to over 200 patients with melanoma.
* This study will use chemotherapy to prepare the immune system before this white blood cell treatment. Our prior studies indicate that aldesleukin may not be required for cell transfer.

Objectives:

- To see if chemotherapy and white blood cell therapy without aldesleukin is a safe and effective treatment for metastatic melanoma.

Eligibility:

- Individuals at least 18 years of age and less than or equal to 70 years of age with metastatic melanoma.

Design:

* Work up stage: Patients will be seen as an outpatient at the National Institute of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed.
* Surgery: If the patients meet all of the requirements for the study they will undergo surgery to remove a tumor that can be used to grow the TIL product.
* Leukapheresis: Patients may undergo leukapheresis to obtain additional white blood cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the TIL cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.
* Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits will take up to 2 days.

DETAILED DESCRIPTION:
BACKGROUND:

- Tumor Infiltrating Lymphocytes (TIL) can mediate the regression of bulky metastatic melanoma when administered to the autologous patient along with high-dose aldesleukin

(IL-2) following a non-myeloablative lymphodepleting chemotherapy preparative regimen.

* IL-2 administration has been shown to increase the number of T regulatory cells and in our trials we have found a direct relationship between the number of IL-2 doses and the reconstitution of patients at one week with cluster of differentiation 4 + forkhead box P3 (CD4+ Foxp3) + T regulatory cells.
* In our analysis of factors that relate to the ability of this treatment to mediate objective responses, we have found a highly significant inverse correlation between reconstitution of CD4+ Foxp3+ T regulatory cells and the likelihood of achieving an objective response.
* In our prior clinical trials of cell transfer using TIL after lymphodepletion with or without

  2 (gray)Gy total body irradiation, patients who experienced an objective response received fewer doses of IL-2 compared to non-responders (p=0.007 and 0.03 respectively).
* High levels of the homeostatic T cell growth factor, IL-15, are present in patient serum after the lymphodepleting regimen at the time of cell transfer.
* These factors raise the possibility that IL-2 administration is not required after cell transfer.

OBJECTIVES:

* The primary objective of this trial is to determine whether objective responses can be mediated in patients with metastatic melanoma who have received a lymphodepleting chemotherapy regimen and adoptive transfer of young tumor infiltrating lymphocytes and no IL-2 administration.
* The secondary objective involves the determination of the level of transferred cells in the blood that persist at about 1 week and 1 month after transfer.

ELIGIBILITY:

* Patients greater than or equal to 18 years old with pathologically confirmed diagnosis of metastatic melanoma.
* Patients with measurable disease, absolute neutrophil count greater than 1000/mm(3) and platelet count greater than 100,000/mm(3).
* Patients not eligible to receive IL-2.

DESIGN:

* Patients with metastatic melanoma will undergo resection to obtain tumor for generation of autologous TIL cultures.
* Patients will receive a non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of young

autologous TIL.

- Patients will be evaluated for objective clinical response and for persistence of the transferred cells.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Measurable metastatic melanoma with available autologous tumor infiltrating lymphocytes (TIL).
* Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
* Greater than or equal to 18 years of age and less than or equal to 70 years of age.
* Able to understand and sign the Informed Consent Document
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Life expectancy of greater than three months
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the treatment.
* Serology:
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription-polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
* Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
* Hematology
* Absolute neutrophil count greater than 1000/mm(3) without the support of filgrastim
* White blood cell (WBC) greater than or equal to 3000/mm(3)
* Platelet count greater than or equal to 100,000/mm(3)
* Hemoglobin > 8.0 g/dl
* Chemistry:
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to to 2.5 times the upper limit of normal
* Serum Creatinine less than or equal to to 1.6 mg/dl
* Total bilirubin less than or equal to to 1.5 mg/dl, except in patients with Gilberts Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria.

* Six weeks must have elapsed since any prior antibody therapy including anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) antibody therapy that could affect any anti-cancer immune response, at the time the patient receives the preparative regimen to allow antibody levels to decline. NOTE: patients who have previously received ipilimumab and have documented gastrointestinal (GI) toxicity must have a colonoscopy with normal colonic biopsies.)
* Patients must be ineligible to receive interleukin-2 (IL-2) based on evidence that may include ischemic heart disease, or arrhythmias, or poor ventricular ejection fraction (< 50%), or respiratory compromise (forced expiratory volume in 1 second (FEV1) < 60%), or clinically significant patient history which in the judgment of the investigator would compromise the patients ability to tolerate aldesleukin.

EXCLUSION CRITERIA:

* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Concurrent systemic steroid therapy.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Patients with a ventricular ejection fraction (less than or equal to 30%), or respiratory compromise (FEV1 less than or equal to 40%).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gogas HJ, Kirkwood JM, Sondak VK. Chemotherapy for metastatic melanoma: time for a change? Cancer. 2007 Feb 1;109(3):455-64. doi: 10.1002/cncr.22427. PMID 17200963
- [Background] Atkins MB, Lotze MT, Dutcher JP, Fisher RI, Weiss G, Margolin K, Abrams J, Sznol M, Parkinson D, Hawkins M, Paradise C, Kunkel L, Rosenberg SA. High-dose recombinant interleukin 2 therapy for patients with metastatic melanoma: analysis of 270 patients treated between 1985 and 1993. J Clin Oncol. 1999 Jul;17(7):2105-16. doi: 10.1200/JCO.1999.17.7.2105. PMID 10561265
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035

RESULTS

PARTICIPANT FLOW:
Groups:
- Immunotherapy for Metastatic Melanoma: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of:
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: Fludarabine 25 mg/m2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Young Tumor Infiltrating Lymphocytes (TIL): Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of young TIL. On day 0, cells (1x10e9 to 2x10e11) will be infused intravenously (i.v.) on the Patient Care Unit over 20 to 30 minutes (between one and four days after the last dose of fludarabine).
Period: Overall Study
Arm/Group | Immunotherapy for Metastatic Melanoma
Started | 18
Completed | 16
Not Completed | 2
Not completed — Death during treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Immunotherapy for Metastatic Melanoma
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response in Patients With Metastatic Melanoma
Description: Response is determined by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: Approximately 2 Years
Measure: Number; unit: participants
Arm/Group | Immunotherapy for Metastatic Melanoma
Number analyzed (Participants) | 18
participants
  Not Evaluable | 1
  Progressive Disease | 12
  Partial Response | 5

2. Secondary Outcome: Level of Persistence of the Transferred Cells in Blood
Description: Determine level of transferred cells in the blood following a non-myeloablative lymphodepleting chemotherapy preparative regimen.
Time Frame: Once week and one month after transfer
Population: No data was collected or analyzed, thus we did not perform an evaluation of persistence for this trial. The reason is that we did not accrue a sufficient number of patients in a timely manner. A minimum of 35 subjects was needed to perform an analysis.
Arm/Group | Immunotherapy for Metastatic Melanoma
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Immunotherapy for Metastatic Melanoma
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy for Metastatic Melanoma (N=18)
Death not associated with CTCAE term (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy for Metastatic Melanoma (N=18)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 6 (6)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 18 (18)
Lymphopenia (Blood and lymphatic system disorders) | 18 (18)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 18 (18)
Platelets (Blood and lymphatic system disorders) | 15 (15)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0x10e9/L) (General disorders) | 1 (1)
Rigors/chills (General disorders) | 2 (2)
Weight gain (General disorders) | 1 (1)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 11 (11) — fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever >38.5 degrees C)
Infection (Infections and infestations) | 6 (6)
ALT/SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1)
Pain (General disorders) | 5 (5)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - Other (Oliguria) (Renal and urinary disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was closed prematurely due to slow and insufficient accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No